CLINICAL TRIAL: NCT02055885
Title: Does Correction of Exercice-induced Desaturation by O2 Improve Systematically Exercise Tolerance in COPD Patients ?
Brief Title: Correction of Exercise-induced Desaturation by Acute Oxygen Supply and Exercise Responses in COPD
Acronym: RePox-1
Status: Completed | Type: Observational
Sponsor: 5 Santé (Other)
Responsible Party: Sponsor
Other Study IDs: Fvie_RePox-1
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Obstructive Pulmonary Disease; Oxygen/Therapeutic Use
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Positive responders: Positive responders (R+): patients exhibiting an increase in the 6WT distance ≥ 10% and/or a decrease in dyspnea ≥ 10% (i.e., ≥ 1 point on the visual analogue scale).
- negative responders: Negative responders(R-): patients exhibiting a decrease in the distance ≥ 10% and/or an increase in dyspnea ≥ 10%.

SUMMARY:
In the literature, the effects of acute oxygen administration on exercise tolerance and related symptoms have often appeared to be contradictory. Some investigations have reported benefits from acute oxygen supply during exertion, including increased exercise performance, reduced dyspnea, and better cardiorespiratory adaptations, whereas other studies have reported no improvement. Recently, we advanced then the hypothesis that some patients would be non-responders and even worsen under oxygen treatment. The preliminary results confirmed our hypothesis since we demonstrated that while 56% of the patients were improved with supplemental oxygen, 16% were non-responders and 28% were negative-responders (decreased performance and increased dyspnea during endurance exercise with supplemental oxygen). However, this was a pilot study offering preliminary insights and tentative conclusions that must be confirmed in a larger case series.

The aims of this retrospective study was :

1. To confirm on cohorte and with clinical test (the 6-minute walking test - 6WT) the deleterious responses to acute oxygen supplementation in LTOT (long terme oxygenotherapy treatment) and non-LTOT patients who exhibit exercise desaturation.
2. To identify the predictive factors among the clinical data (i.e., anthropometric, spirometric and gazometric data) and/or functional data recorded during rehabilitation program

DETAILED DESCRIPTION:
During this study, a retrospective data collection will be carried out using the informations contained in the medical folders of patients admitted in our centers for pulmonary rehabiliation program.

We will select patients who meet the following criteria:

A) patients having two 6WT early in their program B) who desaturate (SpO2 <90% for 3 consecutive min) during the first 6WT and who will have been properly corrected with a supply of oxygen during the second walk test.

The analyzed parameters will be distance and dyspnea during the tests

ELIGIBILITY:
Inclusion Criteria:

* Obstructive airflow limitation defined by FEV1/CVF < 70% and FEV1 < 80 %
* Patients with or without long terme oxygenotherapy
* Patients exhibited during the first test, an exercise-induced desaturation, defined by SaO2 < 90% for 3 consecutive minutes during the 6-minute walking test in the air condition for non-LTOT or with the flow normally recommended during exercise for LTOT patients (i.e., flow rate of rest + 1L/min)
* Patients with no desaturation during the test with oxygen supply

Exclusion Criteria:

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic obstructive pulmonary disease and exhibiting an exercise-induced desaturation during six minute walkink test.
Sampling Method: Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2014-02; Primary Completion 2014-02 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Distance of six minute walking test (meter) | Baseline

SECONDARY OUTCOMES:
Dyspnea during the 6 minute walking test | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nelly N HERAUD, Pd-D, Study Director — 5 Santé
Locations (2):
- France (2):
  - Clinique du Souffle La Vallonie, Lodève
  - Clinique du Souffle La Solane, Osséjà

REFERENCES:
- [Background] Heraud N, Prefaut C, Durand F, Varray A. Does correction of exercise-induced desaturation by O(2) always improve exercise tolerance in COPD? A preliminary study. Respir Med. 2008 Sep;102(9):1276-86. doi: 10.1016/j.rmed.2008.04.005. Epub 2008 Jul 10. PMID 18619828